CLINICAL TRIAL: NCT02953769
Title: Use of Prevena Incision Management System in Wound Morbidity in Complex Ventral Hernia Patients. A Prospective Randomized Control Trial
Brief Title: Prevena Incision Management System Wound Care
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator left the Hospital and did not transfer the study
Sponsor: AdventHealth (Other)
Collaborators: KCI USA, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: 951279
Record Dates: First submitted 2016-11-01; First posted 2016-11-03 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Arm 1: Ventral hernia repair using standard wound care.
- Arm 2: Ventral hernia repair, regarding wound morbidity, post-operative pain and patient comfort to ambulation, with the use of Prevena™

SUMMARY:
Comparison of ventral hernia repair using standard wound care versus Prevena.

DETAILED DESCRIPTION:
Compare the outcomes for patients who have abdominal reconstruction for ventral hernia repair, regarding wound morbidity, post-operative pain and patient comfort to ambulation, with the use of Prevena™ to those patients who have ventral hernia repair to those who have standard wound care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 - 89
2. Open ventral hernia repair with or abdominal wall reconstruction after midline or non-midline defects.
3. Able to provide informed consent

Exclusion Criteria:

1. Immunosuppresses patients
2. Children 0 - 17

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Elective Ventral hernia repair
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-10-16 (Actual); Study Completion 2018-10-16 (Actual)

PRIMARY OUTCOMES:
Primary Objective for Wound Care Comparison | December 31, 2017
  To quantify differences in the routine care of wound morbidity versus the use of Prevena™ by observing the healing process and obtaining quality of life by using the Carolinas Comfort Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Parra Davila, MD, Principal Investigator — Physician
Locations (1):
- Florida Hospital Celebration Health, Celebration, Florida, United States

IPD SHARING:
Plan to Share IPD: No